CLINICAL TRIAL: NCT07013058
Title: Evaluation of the Efficacy of a Nigella Sativa Extract Standardized to 10% Thymoquinone (Nisatol®) in Improving Metabolic and Blood Pressure Parameters and Quality of Life in Perimenopausal Women With Metabolic Syndrome: A Prospective, Multicenter, Randomized Controlled Clinical Trial
Brief Title: Evaluation of a Nigella Sativa Extract (10% Thymoquinone, Nisatol®) in Perimenopausal Women With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Collaborators: University of Urbino "Carlo Bo" (Other)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor of Clinical Biochemistry and Experimental medicine, Liaquat University of Medical & Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 134_21May2025_NISATOL
Record Dates: First submitted 2025-05-29; First posted 2025-06-10 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Metabolic Syndrome; Elevated Blood Pressure
MeSH Terms: conditions — Metabolic Syndrome; Hypertension | interventions — Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to receive either Nisatol® (Nigella sativa extract) or follow a Mediterranean diet for 4 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nisatol® Supplement Group (Experimental): Participants in this arm will receive 2 softgel capsules per day of Nigella sativa oil standardized to 10% thymoquinone (Nisatol®), one capsule with lunch and one with dinner, for a total duration of 4 months.
  Interventions: Dietary Supplement: Nigella sativa extract (Nisatol®)
- Mediterranean Diet Group (Active Comparator): Participants in this arm will follow a Mediterranean diet for 4 months. No Nigella sativa supplement will be administered.
  Interventions: Behavioral: Mediterranean Diet

INTERVENTIONS:
Dietary Supplement: Nigella sativa extract (Nisatol®) — Participants will take 2 softgel capsules daily of Nigella sativa oil standardized to 10% thymoquinone (Nisatol®), one capsule with lunch and one with dinner, for 4 months.
  Arms: Nisatol® Supplement Group
Behavioral: Mediterranean Diet — Participants will follow a Mediterranean diet for 4 months under dietary guidance, without receiving any Nigella sativa supplementation.
  Arms: Mediterranean Diet Group

SUMMARY:
A prospective, multicenter, randomized controlled study evaluating the efficacy and safety of a Nigella sativa extract standardized to 10% thymoquinone (Nisatol®) in perimenopausal women with metabolic syndrome. The study will assess changes in metabolic and blood pressure parameters, as well as improvements in menopausal symptoms and quality of life.

DETAILED DESCRIPTION:
This prospective, multicenter, randomized controlled clinical trial aims to evaluate the efficacy and safety of a food supplement containing Nigella sativa oil standardized to 10% thymoquinone (Nisatol®) in perimenopausal women diagnosed with metabolic syndrome and experiencing climacteric symptoms.

Fifty participants will be randomly assigned to either the intervention group (receiving 2 softgel capsules of Nisatol® daily for 4 months) or a control group following a Mediterranean diet. The primary endpoint is the change from baseline in metabolic and blood pressure parameters, including fasting glucose, lipid profile, cortisolemia, uricemia, and systolic/diastolic blood pressure. The study will also assess quality of life using the Greene Climacteric Scale and monitor treatment safety and tolerability.

The study addresses the need for non-hormonal, evidence-based interventions for managing metabolic and menopausal symptoms in midlife women.

ELIGIBILITY:
Inclusion Criteria:

* Perimenopausal women aged 40-60 years
* Presence of climacteric (menopausal) symptoms
* Diagnosis of metabolic syndrome, defined as alteration of at least 3 of the following:

  * Systolic blood pressure ≥130 mmHg and/or diastolic ≥85 mmHg
  * HDL cholesterol <50 mg/dL
  * Triglycerides ≥150 mg/dL
  * Fasting blood glucose ≥100 mg/dL
  * Uricemia >7 mg/dL

Exclusion Criteria:

* Use of hormone replacement therapy (HRT)
* Presence of neoplastic diseases
* Presence of liver disease, kidney failure, or diabetes mellitus
* Drug or alcohol abuse
* Known hypersensitivity to Nigella sativa or any formulation component

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2025-06-15 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
Change in Fasting Blood Glucose | Baseline to 4 months
  Evaluation of the change in fasting blood glucose from baseline to 4 months.
Change in Total Cholesterol levels, (mg/dL) | Baseline to 4 months
  Evaluation of total cholesterol from baseline to 4 months.
Change in low-density lipoprotein cholesterol levels, (mg/dL) | Baseline to 4 months
  Evaluation of low-density lipoprotein cholesterol from baseline to 4 months.
Change in high-density lipoprotein cholesterol levels, (mg/dL) | Baseline to 4 months
  Evaluation of high-density lipoprotein cholesterol from baseline to 4 months.
Change in Triglycerides levels, (mg/dL) | Baseline to 4 months
  Evaluation of triglyceride levels from baseline to 4 months.
Change in Blood Pressure | Baseline to 4 months
  Evaluation of the change in systolic and diastolic blood pressure from baseline to 4 months.
Change in Serum Cortisol levels, (μg/dL) | Baseline to 4 months
  Evaluation of Cortisol levels from baseline to 4 months.
Change in Serum Uric Acid levels, (mg/dL) | Baseline to 4 months
  Evaluation of Uric acid levels from baseline to 4 months.
Change in serum Alanine Aminotransferase Enzyme levels, (U/L) | Baseline to 4 months
  Evaluation of Alanine Aminotransferase Enzyme levels from baseline to 4 months.
Change in serum Aspartate Aminotransferase Enzyme levels, (U/L) | Baseline to 4 months
  Evaluation of Aspartate Aminotransferase Enzyme levels from baseline to 4 months.
Change in serum Change in Serum Creatinine levels, (mg/dL or µmol/L) | Baseline to 4 months
  Evaluation of serum creatinine from baseline to 4 months.
Change in serum Creatine Phosphokinase Enzymes levels, (U/L) | Baseline to 4 months
  Evaluation of Creatine Phosphokinase Enzymes levels from baseline to 4 months.
Change in Climacteric Symptoms | Baseline to 4 months
  Evaluation using the Greene Climacteric Scale, a 21-item self-reported questionnaire where each item is rated from 0 (not at all) to 3 (extremely), with a total score range from 0 to 63. Higher scores indicate more severe symptoms. Changes will be measured from baseline to 4 months.

SECONDARY OUTCOMES:
Safety and Tolerability | Throughout study duration (4 months)
  Evaluation of adverse events, tolerability score (0-10), and adherence rate (%) over the 4-month treatment period.

CONTACTS AND LOCATIONS:
Locations (1):
- ASL Frosinone, Dipartimento di Prevenzione,, Frosinone, Italy

IPD SHARING:
Plan to Share IPD: No